CLINICAL TRIAL: NCT05085561
Title: A Two-Part Study of REC-994 in the Treatment of Adults With Symptomatic Cerebral Cavernous Malformation (CCM); Part 1: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Safety, Efficacy and Pharmacokinetics of Two Doses of REC-994; Part 2: A Long-Term Blinded Extension Clinical Trial to Evaluate Long-Term Safety Tolerability and Efficacy of REC-994
Brief Title: The Symptomatic Cerebral Cavernous Malformation Trial of REC-994
Acronym: SYCAMORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Recursion Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC-994-201
Record Dates: First submitted 2021-10-08; First posted 2021-10-20 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Cavernous Malformation
Keywords: Cerebral Cavernous Malformation; CCM
MeSH Terms: conditions — Hemangioma, Cavernous, Central Nervous System

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- REC-994 200 mg (Active Comparator): REC-994 200 mg po once daily (QD) (1 200 mg REC-994 tablet, 1 matching placebo tablet)
  Interventions: Drug: REC-994; Drug: Placebo
- REC-994 400 mg (Active Comparator): REC-994 400 mg po QD (2 200 mg REC-994 tablets)
  Interventions: Drug: REC-994
- Placebo (Placebo Comparator): Matching Placebo po QD (2 matching placebo tablets)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REC-994 — REC-994 200 mg tablets
  Arms: REC-994 200 mg; REC-994 400 mg
Drug: Placebo — Placebo Tablets
  Arms: Placebo; REC-994 200 mg

SUMMARY:
This is a two-part, multi-center, randomized, double-blind, placebo-controlled study to investigate the safety, efficacy and pharmacokinetics of REC-994 (200 mg and 400 mg) compared to placebo in participants with symptomatic cerebral cavernous malformation (CCM).

DETAILED DESCRIPTION:
Part 1: Participants will receive treatment over a period of 12 months. Part 2: Optional long-term extension (LTE) for participants completing Part 1 and who are eligible for extended treatment with REC-994.

ELIGIBILITY:
Inclusion criteria:

1. 18 years of age or older with anatomic CCM lesions demonstrated by brain MRI
2. Have symptomatic CCM
3. Have provided written informed consent to participate in the study
4. Have not participated in a clinical trial utilizing an investigational agent within 28 days or within 5 half-lives of the investigational drug (whichever is longer) prior to Screening

Exclusion Criteria:

1. Symptoms deemed by the study Investigator to be caused exclusively by irreversible neuronal damage from prior stroke or neurosurgical instrumentation
2. History of cranial irradiation or surgical/radiosurgical treatment of the primary symptomatic CCM lesion
3. Pregnant or breast feeding
4. Be unable or unwilling to participate in MRI assessments (e.g., claustrophobia, metal implant or implanted cardiac pacemaker)
5. Liver dysfunction or active liver disease as defined by baseline serum transaminases >2x upper limit of normal (ULN)
6. Have moderately or severely impaired renal function (estimated glomerular filtration rate [eGFR] <60ml/min) or active renal disease or have previously received a kidney transplant
7. Have had a previous diagnosis of skeletal muscle disorders (myopathy) of any cause or have a baseline creatine kinase level > 5x ULN
8. History of alcohol or substance abuse within 1 year prior to screening
9. Clinically significant laboratory abnormality
10. Have had an intracerebral hemorrhage within 3 months of screening or any brain surgery within 6 months of screening (not including the primary symptomatic CCM lesion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Up to 24 months

SECONDARY OUTCOMES:
Change in patient reported outcomes (Cerebral Cavernous Malformation Health Index) | Up to 24 months
Change in patient reported outcomes (Modified Rankin Scale) | Up to 24 months
Change in patient reported outcomes (SymptoMScreen Score) | Up to 24 months
Change in disease-associated symptoms (number of MRI-confirmed cerebral hemorrhagic events) | Up to 24 months
Plasma concentrations of REC-994 | Up to 12 months

OTHER OUTCOMES:
Change in disease-associated symptoms (size and number of lesions on MRI) | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Xenoscience Inc, Phoenix, Arizona
  - UCLA, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Florida, Gainesville, Florida
  - Lyerly Neurosurgery, Jacksonville, Florida
  - Cleveland Clinic Florida, Port Saint Lucie, Florida
  - Emory, Atlanta, Georgia
  - Valley Hospital, Ridgewood, New Jersey
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No